CLINICAL TRIAL: NCT05708404
Title: A Novel Outpatient Treatment for Patients With Severe and Enduring Anorexia Nervosa: Patient Characteristics, Treatment Goals, and Course of Treatment.
Brief Title: Outpatient Treatment of Severe and Enduring Anorexia Nervosa
Status: Completed | Type: Observational
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Monica Algars, Ph.D., Helsinki University Central Hospital
Other Study IDs: PISARAAVO
Record Dates: First submitted 2023-01-11; First posted 2023-02-01 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Anorexia
Keywords: Anorexia nervosa; Severe and enduring anorexia nervosa; Treatment
MeSH Terms: conditions — Anorexia; Anorexia Nervosa

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Outpatient treatment of severe and enduring anorexia nervosa — A novel outpatient treatment of severe and enduring anorexia nervosa, aiming at enhancing quality of life and minimizing harm

SUMMARY:
Approximately 20-30 % of individuals with the eating disorder anorexia nervosa develop an enduring form of the illness. In this study a new treatment for patients with severe and enduring anorexia nervosa was described. The treatment is flexible and aims at enhancing quality of life. The participants consisted of all referrals resulting in an assessment or treatment period at the unit between May 2017 and May 2022. The study was a registry study. Information regarding patient characteristics, treatment goals, and the course of treatment was gathered from medical records.

ELIGIBILITY:
Inclusion criteria:

* Age ≥ 18 years
* A referral resulting in an assessment or treatment period at the unit for patients with severe and enduring anorexia nervosa at the HUS Helsinki University Hospital between May 2017 and May 2022.

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Adult women with severe and enduring anorexia nervosa.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
How the treatment goals were met | At the end of treatment, an average of 15.4 months
  Whether or not the patients' individual treatment goals, defined at the beginning of treatment, had been met, partly met, or not met at the end of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Jaana Suokas, Ph.D., Principal Investigator — HUS Helsinki Central Hospital
Locations (1):
- HUS Syömishäiriöyksikkö, Helsinki, PL 282, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Algars M, Oshukova S, Suokas J. A novel outpatient treatment model for patients with severe and enduring anorexia nervosa: an observational study of patient characteristics, treatment goals, and treatment course. J Eat Disord. 2023 Sep 6;11(1):150. doi: 10.1186/s40337-023-00877-x. PMID 37674214